CLINICAL TRIAL: NCT06219044
Title: Ovarian Reserve, Recurrence Rate and Histopathologic Evaluation After DWLS Diode Laser Vaporization of Ovarian Endometriomas: Results From a Prospective, Multicentre, Clinical Trial.
Brief Title: Evaluation of Ovarian Reserve and Recurrence Rate After DWLS Diode Laser OMA Vaporization
Acronym: OMAlaser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Collaborators: University of Foggia (Other); Azienda Ospedaliera per l'Emergenza Canizzaro (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Full Professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMA Diode Laser Vaporization
Record Dates: First submitted 2023-12-23; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Endometrioma; Ovarian Endometriosis; Ovarian Endometrioma
Keywords: endometrioma; laparoscopy; diode laser
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- symptomatic ovarian endometrioma (Experimental): patients aged between 18 and 40 years with clinical and/or ultrasound diagnosis of symptomatic ovarian endometrioma
  Interventions: Procedure: laparoscopic endometrioma laser vaporization

INTERVENTIONS:
Procedure: laparoscopic endometrioma laser vaporization — laser vaporization of ovarian endometrioma using a DWLS diode laser during a laparoscopy

SUMMARY:
PURPOSE OF THE STUDY The study aims to evaluate the effectiveness of the Dual Wavelength Laser System (DWLS) diode laser on the treatment of endometrioma (OMA), with ablation and vaporization of the cystic capsule without performing the stripping technique, in terms of ovarian reserve and recurrence rate.

DETAILED DESCRIPTION:
BACKGROUND Endometriosis cyst, or endometrioma (OMA), is one of the most frequent gynaecological pathologies and is commonly associated with symptoms such as infertility and chronic pelvic pain. Randomized and meta-analysis studies demonstrate how the most effective surgery, in terms of percentages of pregnancy after surgery and minor rates of recurrence of cysts or pelvic pain, is the complete removal of the cyst wall through laparoscopic "stripping". However, data has recently emerged on the possible damage determined by "stripping" surgery on the healthy ovarian tissue adjacent to the OMA.

Studies on the anatomopathological characteristics of the wall of the OMA surgically removed have shown that, with the complete removal surgery, part of ovarian tissue is inadvertently removed together with the OMA wall in almost all cases since there is no real cleavage plan between cysts and healthy ovarian tissue. The post-surgery ovarian reserve has been reported, measured as lower levels of antimullerian hormone (AMH), minor values of antral follicular count (AFC), and reduced postoperative ovarian volumes. Worst performances have also been reported for the induction of ovulation for in vitro fertilization techniques. In the event of the removal of bilateral OMA, 2-4% of early premature ovarian failure has been reported, confirming possible surgical damage to healthy ovarian tissue. Following these data, the international scientific community has begun to question the effective superiority of the complete removal approach of the cystic wall, or "stripping", given these new acquisitions on post-surgical ovarian damage. Therefore, the theme of the best therapeutic approach to OMA has become one of the most debated in the gynaecological field. Despite the data on the possible surgical damage, surgical intervention remains one of the cornerstones of OMA therapy.

The recurrence rate evaluation is one of the primary endpoints of all OMA surgery studies. Guo S.w. has estimated a recurrence rate of 21.5% to 2 years and 40-50% to 5 years. In a recent systematic review of Ceccaroni M. et al., 12-30% recurrence rates are shown 2-5 years after surgical treatment.

An alternative technique to "stripping" is the fenestration of the cyst followed by ablation or vaporization with the laser of the internal wall of the cyst left "in situ" without the complete removal of the cystic wall with healthy ovarian tissue. Candiani et al. demonstrated, in their randomized study, that the "One Step" vaporization of the OMA capsule with the CO2 laser is more effective than stripping in reducing the residual follicular damage (in terms of AMH and AFC).

For better results regarding controlled ablation of the cystic wall of the OMA, the DWLS diode laser could be helpful. The combination of two wavelengths, 980 Nm and 1470 Nm, gives a contemporary absorption in H2O and haemoglobin with an excellent ability of hemostasis, cut and vaporization, as previously demonstrated in laparoscopic and hysteroscopic surgery.

PURPOSE OF THE STUDY The study aims to evaluate the effectiveness of the DWLS diode laser on the treatment of OMA, with ablation and vaporization of the cystic capsule without performing the stripping technique, in terms of ovarian reserve, recurrence rate and patient's symptoms.

Primary objective Evaluation of the ovarian reserve regarding AFC, AMH and the patient's symptoms.

Secondary objective Evaluation of OMA recurrence rates on the treated ovary and pregnancy rate of the patients operated on.

EXPECTED BENEFITS Compared to the stripping technique with complete removal of the cystic wall, this approach could make the treatment easier and faster but, above all, less harmful for the healthy ovarian parenchyma below the cyst.

Compared to the one-step technique with CO2 laser, the combination of the two wavelengths of diode lasers would allow a more controlled ablation of the endometriosis tissue for its well-known characteristics of hemostasis and vaporization even in the most bloody tissues e irrigated by physiological solution.

INTERVENTION STRATEGY AND INSTRUMENTS The investigators plan to recruit 70 patients of reproductive age with mono of bilateral OMA with a diameter ≥ 3 and ≤ 8 cm associated with infertility or pelvic pain who have never carried out previous interventions on one or both annexes. The cyst diameter cut-offs were chosen according to the previous data present in the literature and guidelines for the management of OMA. The patients will be evaluated at the endometriosis/chronic pelvic pain centre of the gynaecology unit of the University Hospital of Monserrato (Cagliari) and in the other centres involved in the study. All patients will perform a visit, a transvaginal ultrasound and where magnetic resonance imaging of the pelvis is necessary to provide accurate information on the location of the endometriosis pathology and to exclude other coexisting uterine or annexial diseases.

All surgical procedures will be performed in operating laparoscopy under general anaesthesia.

In all patients, the diagnosis of OMA will be confirmed by surgical exploration and histopathological examination.

During the surgery, the DWLS diose laser will be used to vaporise the endometrioma capsule after opening, aspiration of the liquid and subversion of the internal wall of the cyst. Before using the laser, an accurate exploration of the cyst capsule and a biopsy on it will be performed. The removed samples will be sent for histological examination by requiring the measurement of the thickness of the endometriosis capsule. After surgery, all patients will be followed over time at quarterly intervals in the first year. At each follow-up visit, the presence of pain symptoms will be checked (dysmenorrhea, dyspareunia, chronic pelvic pain, dyschezia, dysuria) in patients operated for pelvic pain and the presence of pregnancy in patients operated by infertility to evaluate the cure or recurrence rates of the symptoms.

Transvaginal ultrasounds will be performed on each control for the evaluation of the presence or absence of a recurrence of OMA. The cyst must have a diameter of at least 2 cm to satisfy the ultrasound criteria for the recurrence of OMA, and it must persist over time (for at least two consecutive menstrual cycles) to be distinguished as a functional cyst.

The AFC will also be assessed During the ultrasound examination between the second and seventh day of the cycle. The AMH will systematically be evaluated for the measurement of the ovarian reserve.

During the first visit, it will be detected:

* Clinical and surgical history
* Full target examination
* Gynecological examination
* Concomitant drugs and their indication
* Pelvic and trans-vaginal ultrasounds were performed between the second and seventh day of the cycle with an evaluation of the parameters of ovarian functionality, OMA volumes, and the ovary and AFC on both ovaries.
* Dosage of the AMH hormone

Follow up evaluation

With quarterly frequency in the first year:

* Clinical evaluation
* Pelvic and trans-vaginal ultrasounds were performed between the second and seventh day of the cycle to evaluate the parameters of ovarian functionality and AFC on both ovaries and possible recurrence of the OMA.
* Dosage of the AMH hormone.

POPULATION Seventy patients aged between 18 and 40 with clinical and ultrasound diagnoses of mono or bilateral OMA cysts. To be suitable for inclusion, patients with an ultrasound diagnosis of mono or bilateral OMA should present symptoms such as pelvic pain or sterility.

STATISTICAL ANALYSIS The data will be tabulated on a specific database and analyzed using specific software. A descriptive output will be created, and the comparison between variables will be made through parametric and non-parametric tests with a level of significance of 95%. The IBM SPSS Statistics software will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years old
* OMA mono or bilateral ≥ 3 and ≤ 8 cm in diameter
* presence of symptoms such as pelvic pain and sterility

Exclusion Criteria:

* Patients who are unable to provide written informed consent or to follow the procedures provided for by the protocol
* Age <18 years and> 40 years
* OMA mono or bilateral <3 and> 8 cm in diameter
* Asymptomatic patients
* Absence of histological confirmation of endometriosis cysts
* previous interventions on one or both annexes
* Failure to follow-up

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — ovarian endometrioma
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the ovarian reserve using AntiMullerian Hormone (AMH) assessment. | every 3 months for one year
  Blood dosage of AntiMullerian Hormone expressed in nanograms/milliliter (ng/mL)
Evaluation of the ovarian reserve using Antral follicular Count (AFC) | every 3 months for one year
  counts of the number of antral follicles present in the ovary during ultrasound scan. The count is presented in Numbers from 0 to any numbers (n°)
Evaluation of the patients' symptoms | every 3 months for one year
  assessed using the Visual Analogue Scale (VAS) , from 0 as the minimum to 10 as maximum value. Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Evaluation of endometrioma recurrence rate | every 3 months for one year
  Ultrasound scan Evaluation of OMA recurrence. Assessed using a percentage (%) of patients who present the endometrioma in the ovaries after surgery
Evaluation of pregnancy rate | every 3 months for one year
  Assessed as percentage (%) of patients who achieved pregnancy after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari,Obstetrics and Gynecological Department, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kennedy S, Bergqvist A, Chapron C, D'Hooghe T, Dunselman G, Greb R, Hummelshoj L, Prentice A, Saridogan E; ESHRE Special Interest Group for Endometriosis and Endometrium Guideline Development Group. ESHRE guideline for the diagnosis and treatment of endometriosis. Hum Reprod. 2005 Oct;20(10):2698-704. doi: 10.1093/humrep/dei135. Epub 2005 Jun 24. PMID 15980014
- [Background] Dunselman GA, Vermeulen N, Becker C, Calhaz-Jorge C, D'Hooghe T, De Bie B, Heikinheimo O, Horne AW, Kiesel L, Nap A, Prentice A, Saridogan E, Soriano D, Nelen W; European Society of Human Reproduction and Embryology. ESHRE guideline: management of women with endometriosis. Hum Reprod. 2014 Mar;29(3):400-12. doi: 10.1093/humrep/det457. Epub 2014 Jan 15. PMID 24435778
- [Background] Benschop L, Farquhar C, van der Poel N, Heineman MJ. Interventions for women with endometrioma prior to assisted reproductive technology. Cochrane Database Syst Rev. 2010 Nov 10;2010(11):CD008571. doi: 10.1002/14651858.CD008571.pub2. PMID 21069706
- [Background] Practice Committee of the American Society for Reproductive Medicine. Endometriosis and infertility: a committee opinion. Fertil Steril. 2012 Sep;98(3):591-8. doi: 10.1016/j.fertnstert.2012.05.031. Epub 2012 Jun 15. PMID 22704630
- [Background] Donnez J, Lousse JC, Jadoul P, Donnez O, Squifflet J. Laparoscopic management of endometriomas using a combined technique of excisional (cystectomy) and ablative surgery. Fertil Steril. 2010 Jun;94(1):28-32. doi: 10.1016/j.fertnstert.2009.02.065. Epub 2009 Apr 9. PMID 19361793
- [Background] Tsolakidis D, Pados G, Vavilis D, Athanatos D, Tsalikis T, Giannakou A, Tarlatzis BC. The impact on ovarian reserve after laparoscopic ovarian cystectomy versus three-stage management in patients with endometriomas: a prospective randomized study. Fertil Steril. 2010 Jun;94(1):71-7. doi: 10.1016/j.fertnstert.2009.01.138. Epub 2009 Apr 25. PMID 19393996
- [Background] Muzii L, Bellati F, Bianchi A, Palaia I, Manci N, Zullo MA, Angioli R, Panici PB. Laparoscopic stripping of endometriomas: a randomized trial on different surgical techniques. Part II: pathological results. Hum Reprod. 2005 Jul;20(7):1987-92. doi: 10.1093/humrep/deh851. Epub 2005 Apr 28. PMID 15860498
- [Background] Guo SW. Recurrence of endometriosis and its control. Hum Reprod Update. 2009 Jul-Aug;15(4):441-61. doi: 10.1093/humupd/dmp007. Epub 2009 Mar 11. PMID 19279046
- [Background] Ceccaroni M, Bounous VE, Clarizia R, Mautone D, Mabrouk M. Recurrent endometriosis: a battle against an unknown enemy. Eur J Contracept Reprod Health Care. 2019 Dec;24(6):464-474. doi: 10.1080/13625187.2019.1662391. Epub 2019 Sep 25. PMID 31550940
- [Background] Seo JW, Lee DY, Yoon BK, Choi D. The age-related recurrence of endometrioma after conservative surgery. Eur J Obstet Gynecol Reprod Biol. 2017 Jan;208:81-85. doi: 10.1016/j.ejogrb.2016.11.015. Epub 2016 Nov 16. PMID 27894033
- [Background] Candiani M, Ottolina J, Posadzka E, Ferrari S, Castellano LM, Tandoi I, Pagliardini L, Nocun A, Jach R. Assessment of ovarian reserve after cystectomy versus 'one-step' laser vaporization in the treatment of ovarian endometrioma: a small randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2205-2211. doi: 10.1093/humrep/dey305. PMID 30299482
- [Background] Angioni S, Pontis A, Sorrentino F, Nappi L. Bilateral salpingo-oophorectomy and adhesiolysis with single port access laparoscopy and use of diode laser in a BRCA carrier. Eur J Gynaecol Oncol. 2015;36(4):479-81. PMID 26390708